CLINICAL TRIAL: NCT03391960
Title: A Compliance Improvement Project to Reduce Central Line Associated Blood Stream Infection (CLABSI) Using a Passive Disinfection Device in an Adult Oncological Hospital in Brazil
Brief Title: Passive Disinfection Cap Compliance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: Eurotrials Brasil Consultores Cientificos Ltda (Industry); 3M (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLIN-PROT-ICH-US-05-319980; Study 05-014137 (Other: 3M)
Record Dates: First submitted 2017-12-07; First posted 2018-01-05 (Actual); Results first posted 2022-02-09 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Infection, Hospital
Keywords: CLABSI; Septicemia; Bloodstream infection; Central line associated bloodstream infection; Catheter related bloodstream infection; Intravascular device; Catheter port
MeSH Terms: conditions — Cross Infection; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Disinfecting barrier cap (Other): In the participating wards, disinfecting barrier cap was used on every needless connector used for accessing CVC IV lines.
  Compliance with disinfecting barrier cap was observed weekly.
  Interventions: Device: Passive disinfection device

INTERVENTIONS:
Device: Passive disinfection device — Add use of passive disinfection cap to existing central line needleless connector infection control procedure
  Other Names: Passive disinfecting cap; Disinfecting cap; Curos disinfecting cap; Curos cap

SUMMARY:
Insertion and maintenance of central venous catheter (CVC) lines are common hospital procedures in patients, including those being treated for cancer. CVCs allow clinicians an access point for infusion of fluids, blood sampling, and measurements, decreasing the need for repeated needle sticks to the patient. However, bloodstream infections associated with CVCs (CLABSIs) are a serious complication, leading to significantly longer hospital stays, morbidity, and mortality. Keeping catheter ports disinfected reduces the risk of bloodstream infection; however, consistent and adequate maintenance and disinfection of the line can be difficult.

The purpose of this study is to demonstrate that passive disinfecting caps can provide a patient safety practice that is easy for clinicians to follow, as well as providing easily auditable compliance, which may lead to lower CLABSI rates.

The compliance rate for needleless connector disinfection will be evaluated after implementation of the passive disinfecting cap, and compared to the pre-intervention rate. The CLABSI rates before and after cap implementation will also be compared.

DETAILED DESCRIPTION:
Insertion and maintenance of central venous catheter (CVC) lines are common hospital procedures in patients, including those being treated for cancer. CVCs allow clinicians an access point for infusion of fluids, blood sampling, and measurements, decreasing the need for repeated needle sticks to the patient. However, bloodstream infections associated with CVCs (CLABSIs) are a serious complication, leading to significantly longer hospital stays, morbidity, and mortality. Keeping catheter ports disinfected reduces the risk of bloodstream infection; however, consistent and adequate maintenance and disinfection of the line can be difficult.

The purpose of this study is to demonstrate that passive disinfecting caps can provide a patient safety practice that is easy for clinicians to follow, as well as providing easily auditable compliance, which may lead to lower CLABSI rates.

Compliance is defined as following the protocol for disinfection of the catheter port. In the pre-intervention period, the disinfection protocol will utilize existing institution scrub-the-hub method. Compliance in the pre-intervention period will be determined by survey.

After the pre-intervention period is complete, passive disinfecting devices (caps) will be implemented hospital-wide for any adult patient using CVC ports.

In the intervention period, the disinfection protocol consists of using the disinfecting barrier cap on every needless connector (catheter port) used for accessing CVC IV lines per protocol. Compliance will be measured using observations, according to a schedule to ensure the absence of a shift bias. Observations will contain the number of needless connectors on CVCs with, and the number of needleless connectors without, disinfecting barrier caps attached.

The compliance rate for needleless connector disinfection will be evaluated after implementation of the passive disinfecting cap, and compared to the pre-intervention rate. The CLABSI rates before and after cap implementation will also be compared.

Incidence of CLABSI will be noted from existing aggregate hospital surveillance system data. The incidence, in terms of catheter days, will be recorded for each assigned intervention ward and for intervention ward overall by month, in the six months before the intervention and in the six-month intervention recording period.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to the participant oncologic hospital
* Adult patients in the assigned intervention units during the seven month intervention period who require needleless connectors for CVC IV tubing access.

Exclusion Criteria:

* Adult patients admitted to the participant oncologic hospital during the seven month intervention period that do not require needleless connectors for CVC IV access during their hospital stay.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A Zimerman, MD, Principal Investigator — Irmandade da Santa Casa de Misericordia de Porto Alegre - ISCMPA
Locations (1):
- 3M HealthCare, Maplewood, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be recorded in the study.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No individual patient was recruited into the study.
Units Other Than Participants: Compliance audits
Groups:
- Compliance With Scrub the Hub Protocol: Compliance with scrub the hub protocol was retrospectively measured through a survey from Health care workers who were working in the hospital and used needleless connector
- Compliance With Disinfecting Barrier Cap Ptotocol: In the participating wards, disinfecting barrier cap was used on every needless connector used for accessing CVC IV lines.
  Compliance with disinfecting barrier cap was observed weekly.
Period: Overall Study
Arm/Group | Compliance With Scrub the Hub Protocol | Compliance With Disinfecting Barrier Cap Ptotocol
Started | 165; 0 Compliance audits (Units were not assessed for this Arm/Group. Data was collected from the health care worker surveys for the retrospective study to monitor compliance with the scrub-the-hub protocol (signed informed consent and were enrolled)) | NA; 156 Compliance audits (No individual patient was recruited into the study. Data was collected from the compliance audits to monitor compliance with the disinfecting barrier cap protocol.)
Completed | 165; 0 Compliance audits | NA; 156 Compliance audits (No individual patient was recruited into the study. Data was collected from the compliance audits to monitor compliance with the disinfecting barrier cap protocol.)
Not Completed | 0; 0 Compliance audits | NA; 0 Compliance audits
Not completed — Protocol Violation | 0 | NA

BASELINE CHARACTERISTICS:
Population: Baseline data were not collected for the health care workers. No individual patient was consented in the study.
Groups:
- Not Applicable: During the study, Baseline data were not collected for the health care workers. No individual patient was consented in the study.
Arm/Group | Not Applicable
Number analyzed (Participants) | 0
Age, Customized — Not Available. Baseline data were not collected for the health care workers.
Sex: Female, Male — Measure Description: Not Available. Baseline data were not collected for the health care workers.
Race (NIH/OMB) — Measure Description: Not Available. Baseline data were not collected for the health care workers.
Study-Specific Measure — Measure Description: Not Available. Baseline data were not collected for the health care workers.

OUTCOME MEASURES:

1. Primary Outcome: Disinfecting Barrier Cap Compliance
Description: Compliance to disinfection protocol for central line needleless connectors. Compliance will be measured by periodic audits, where the number of disinfecting caps on central line needleless connectors is compared to the total number of central line needleless connectors to determine compliance percentage.
Time Frame: 6-month prospective period
Population: No patients assessed for disinfecting barrier cap compliance. Compliance with disinfecting barrier cap was measured by observation of numbers of applicable capped, uncapped ports and misused caps. A total of 156 audits were performed.
Measure: Mean (Standard Deviation); unit: percentage of connector with compliance
Units Other Than Participants: Compliance audits
Groups:
- Disinfecting Barrier Cap Compliance: In the participating wards, disinfecting barrier cap was used on every needless connector used for accessing CVC IV lines.
  Compliance with disinfecting barrier cap was observed weekly.
Arm/Group | Disinfecting Barrier Cap Compliance
Number analyzed (Participants) | NA
Number analyzed (Compliance audits) | 156
percentage of connector with compliance | 98.43 (4.18)

2. Primary Outcome: Scrub the Hub Protocol Compliance
Description: Compliance with Scrub the hub protocol
  Data collected retrospectively by survey
Time Frame: 6-month retrospective period
Population: Compliance with scrub the hub was retrospectively obtained by a survey from 165 healthcare workers who were using needlessness connectors for patient IV access. One was excluded from the compliance analysis due to an inconsistency in the survey data. No patients assessed for disinfecting barrier cap compliance.
Measure: Mean (Standard Deviation); unit: percentage of protocol compliance
Groups:
- Scrub the Hub Protocol Compliance: Compliance with Scrub the hub protocol
  Data collected by survey
  No individual patient's information was collected during the study
Arm/Group | Scrub the Hub Protocol Compliance
Number analyzed (Participants) | 164
percentage of protocol compliance | 5.95 (21.36)

3. Secondary Outcome: CLABSI Rate
Description: Central-line associated blood stream infection assessments were performed once a month per ward during the pre-intervention and post-intervention periods. The total number of CLABSI infections and CVC/day were recorded in all assessments to determine the CLABSI rate per 1000 CVC/days.
  Infections from patients without CVC IV access (those using a three-lumen dialysis catheter with a needleless connector on the third lumen and those using two-lumen dialysis catheters) were also recorded as part of the aggregated data, due to the impossibility of separating the infections in these patients from the ones with CVC access
Time Frame: 6-month retrospective period and 6-month prospective period
Population: Patients who require needleless connectors for CVC IV access or dialysis catheters in one ICU (6 units) and five non-ICU (6 units of each) wards. Total 36 units. No individual patients were enrolled in this study. No Patients assessed for this measure.
Measure: Number; unit: CLABSI rate per 1000 catheter days
Units Other Than Participants: ICU and non-ICU wards
Groups:
- CLABSI Rate for Pre-intervention Period: Number of CLABSI infections and CVC/day recorded during 6 pre-intervention months were used to determine the rate of CLABSI during the 6-month pre-intervention period.
- CLABSI Rate for Post-intervention Period: Number of CLABSI infections and CVC/day recorded during prospective period were used to determine the rate of CLABSI during the 6-month post-intervention period.
Arm/Group | CLABSI Rate for Pre-intervention Period | CLABSI Rate for Post-intervention Period
Number analyzed (Participants) | NA | NA
Number analyzed (ICU and non-ICU wards) | 36 | 36
CLABSI rate per 1000 catheter days | 2.9 | 3.2

4. Secondary Outcome: Catheter-associated Urinary Tract Infection (CAUTI) Rate
Description: Rate of CAUTI per 1000 indwelling urinary catheter days. CAUTI data was recorded to control for possible seasonal and/or environmental effects that could also influence CLABSI and hospital infection rates overall. Data on this type of infection was only available for the ICU, as recording of CAUTI is only mandatory in the intensive care setting in Brazil.
Time Frame: 6 months pre-intervention and 6 months post intervention
Population: Infections from patients with indwelling urinary catheters in one ICU ward. Total 6 units. No individual patients were enrolled in this study. No patients assessed for this measure.
Measure: Number; unit: CAUTI rate per 1000 catheter days
Units Other Than Participants: Units in ICU ward
Groups:
- CAUTI Rate 6 Months Pre-intervention: CAUTI rate per 1000 catheter/days during 6 months pre-intervention
- CAUTI Rate 6 Months Post-intervention: CAUTI rate per 1000 catheter/days during 6 months post intervention
Arm/Group | CAUTI Rate 6 Months Pre-intervention | CAUTI Rate 6 Months Post-intervention
Number analyzed (Participants) | NA | NA
Number analyzed (Units in ICU ward) | 6 | 6
CAUTI rate per 1000 catheter days | 0.78 | 2.26

5. Secondary Outcome: Ventilator-associated Pneumonia (VAP) Rate
Description: Rate of VAP per 1000 ventilator days. VAP data was recorded to control for possible seasonal and/or environmental effects that could also influence CLABSI and hospital infection rates overall. Data on this type of infection was only available for the ICU, as recording of VAP is only mandatory in the intensive care setting in Brazil.
Time Frame: 6-month retrospective period and 6-month prospective period
Population: Infections from patients who have been intubated and received mechanical ventilation in one ICU ward (6 units). No Patients assessed for this measure.
Measure: Number; unit: VAP rate per 1000 ventilator days
Units Other Than Participants: Units in ICU ward
Groups:
- VAP Rate Pre-intervention: VAP rate per 1000 ventilator days 6 months pre-intervention
- VAP Rate Post Intervention: VAP rate per 1000 ventilator days 6 months post-intervention
Arm/Group | VAP Rate Pre-intervention | VAP Rate Post Intervention
Number analyzed (Participants) | NA | NA
Number analyzed (Units in ICU ward) | 6 | 6
VAP rate per 1000 ventilator days | 6.2 | 5.35

6. Secondary Outcome: MBI-Related CLABSI Rate
Description: Central-line associated blood stream infection assessments were performed once a month per ward during the pre-intervention and post-intervention periods. The total number of CLABSI infections and CVC/day were recorded in all assessments. Lastly, CLABSIs were divided into mucosal-barrier injury (MBI)-related and non-MBI-related and recorded separately in the eCRF. MBI-related CLABSIs and CVC/day were used to determine MBI CLABSI rate per 1000 CVC/days.
  Infections from patients without CVC IV access (those using a three-lumen dialysis catheter with a needleless connector on the third lumen and those using two-lumen dialysis catheters) were also recorded as part of the aggregated data, due to the impossibility of separating the infections in these patients from the ones with CVC access.
Time Frame: 6-month retrospective period and 6-month prospective period
Population: as for outcome 3
Measure: Number; unit: MBI CLABSI rate per 1000 catheter days
Units Other Than Participants: ICU and non-ICU wards
Groups:
- MBI-related CLABSI Rate for Pre-intervention Period: Number of MBI CLABSI infections and CVC/day recorded during 6 months of pre-intervention were used to determine the rate of MBI CLABSI during the pre-intervention period.
- MBI-related CLABSI Rate for Prospective Period: Number of MBI CLABSI infections and CVC/day recorded during 6 months of prospective period were used to determine the rate of MBI CLABSI during the prospective period.
Arm/Group | MBI-related CLABSI Rate for Pre-intervention Period | MBI-related CLABSI Rate for Prospective Period
Number analyzed (Participants) | NA | NA
Number analyzed (ICU and non-ICU wards) | 36 | 36
MBI CLABSI rate per 1000 catheter days | 1 | 1.28

7. Secondary Outcome: Non MBI-related CLABSI Rate
Description: Central-line associated blood stream infection assessments were performed once a month per ward during the pre-intervention and post-intervention periods. The total number of CLABSI infections and CVC/day were recorded in all assessments. Lastly, CLABSIs were divided into mucosal-barrier injury (MBI)-related and non-MBI-related and recorded separately in the eCRF. Non MBI-related CLABSIs and CVC/day were used to determine Non-MBI CLABSI rate per 1000 CVC/days.
  Infections from patients without CVC IV access (those using a three-lumen dialysis catheter with a needleless connector on the third lumen and those using two-lumen dialysis catheters) were also recorded as part of the aggregated data, due to the impossibility of separating the infections in these patients from the ones with CVC access.
Time Frame: 6-month retrospective period and 6-month prospective period
Population: as for outcome 3
Measure: Number; unit: CLABSI rate per 1000 catheter days
Units Other Than Participants: ICU and non-ICU wards
Groups:
- Non-MBI CLABSI Rate for Pre-intervention Period: Number of Non-MBI CLABSI infections and CVC/day recorded during 6 months of pre-intervention were used to determine the rate of CLABSI during the pre-intervention period
- Non-MBI CLABSI Rate for Prospective Period: Number of Non-MBI CLABSI infections and CVC/day recorded during 6 months of prospective period were used to determine the rate of CLABSI during the prospective period.
Arm/Group | Non-MBI CLABSI Rate for Pre-intervention Period | Non-MBI CLABSI Rate for Prospective Period
Number analyzed (Participants) | NA | NA
Number analyzed (ICU and non-ICU wards) | 36 | 36
CLABSI rate per 1000 catheter days | 1.93 | 1.92

ADVERSE EVENTS:
Time Frame: No individual patient data (including adverse events [AEs]) were recorded during this study.
Description: No individual patient data (including adverse events [AEs]) were recorded during this study as no individual patient was enrolled into the study .
Groups:
- EG000: No individual patient data (including adverse events [AEs]) were recorded during this study.
Arm/Group | EG000
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
The rate of CLABSI per 1000 central line days was determined by using aggregated data on infections and on CVC/day during the study period. Infections from patients without CVC IV access were also part of the aggregated data recorded. However, as these patients did not have CVC access, they did not contribute to the CVC/day data collected throughout the study. As a result, the rate of CLABSI may have been overestimated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT03391960/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/60/NCT03391960/SAP_001.pdf